CLINICAL TRIAL: NCT07167225
Title: Carcinogen and Toxicant Exposure Among Young Adults Who Co-Use E-cigarettes and Cannabis (Co-Tox Study)
Status: Recruiting | Type: Observational
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: I-4235024
Record Dates: First submitted 2025-08-27; First posted 2025-09-11 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Cigarette Smoking-Related Carcinoma; E-Cig Use
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- E-cigarette consumers: Predominant e-cigarette consumers
  Interventions: Other: Effectiveness of different recruitment approaches; Other: Choice of study completion locations; Other: E-cigarette dependence Scale
- Cannabis consumers: Predominant cannabis consumers
  Interventions: Other: Effectiveness of different recruitment approaches; Other: Choice of study completion locations; Other: Cannabis Engagement Assessment
- e-cigarette -cannabis coconsumers: Consumers who use both e-cigarettes and cannabis .
  Interventions: Other: Effectiveness of different recruitment approaches; Other: Choice of study completion locations; Other: Cannabis Engagement Assessment; Other: E-cigarette dependence Scale

INTERVENTIONS:
Other: Effectiveness of different recruitment approaches — Subjects will asked which type of recruitment material they've seen when completing the screening survey
Other: Choice of study completion locations — subjects will choose location when coordinator calls to schedule appointment
Other: Cannabis Engagement Assessment — Self reported measure of current cannabis use that contains 30 questions assessing quantity, frequency of use and method of consumption in the past 30 days.
  Groups: Cannabis consumers; e-cigarette -cannabis coconsumers
Other: E-cigarette dependence Scale — A 22-item questionnaire measuring e-cigarette dependence. Higher scores indicate greater dependence.
  Groups: E-cigarette consumers; e-cigarette -cannabis coconsumers

SUMMARY:
This study evaluates the amount of nicotine, cannabis, and toxicants linked to the use of nicotine e-cigarette and/or cannabis products in the blood and urine of young adult users as well as the cannabis and nicotine use behaviors of consumers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate differences in self-reported nicotine and cannabis use behaviors and biomarkers of exposure to toxicants and carcinogens by product use status, to generate effect sizes required to calculate sample sizes needed for a larger study.

ELIGIBILITY:
Inclusion Criteria:

* Young adult (18-25 years old).
* Ability to read and write in English.
* Participants must fall into one of the following groups (based on self-report):
* Predominant e-cigarette consumer: defined as using nicotine-containing e-cigarettes daily for the past six months but not having used other nicotine containing products more than weekly or cannabis products for the past month.
* Predominant cannabis consumer: defined as using cannabis at least 3x/week for the past six months in any form, including smoking, vaping, and oral use, with no more than weekly use of any nicotine or tobacco products.
* E-cigarette-cannabis co-consumers: defined as daily use of nicotine e-cigarettes and use of cannabis at least 3x/week, including smoking, vaping, and oral use, for at least the past six months, with no use of other nicotine containing products more than weekly.
* No self-reported diagnosis of kidney disease (current, or within the past year prior to the study visit).
* Participants must understand the voluntary nature of this study and sign a written informed consent form before proceeding with study activities.

Exclusion Criteria:

* Individuals under the age of 18 or over the age of 25.
* Currently pregnant or breastfeeding (female participants).
* Unwilling or unable to follow protocol requirements

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young adults (18-25 year old) currently using cannabis products and/or electronic cigarettes containing nicotine.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Differences in biomarker levels across groups | 1 study session lasting 1 hour
  Will compare the mean biomarker levels between groups using a one-way ANOVA model, with Bonferroni-adjusted pairwise comparisons, as appropriate.

SECONDARY OUTCOMES:
Differences in self reported nicotine and cannabis use behaviors | 1 study session (1 hour)
  Self reported questionnaire
Differences in psychosocial characteristics by group | 1 study session (1 hour)
  Will be compared between groups using the appropriate general linear models. All model and test assumptions will be verified graphically, with transformations applied as appropriate.
Study interest | Up to 1 year
  Study interest and eligibility Measured via number of contacts to inquire about the study, and number of eligible applicants. The eligibility and interest rates of the individuals approached and the completion rates of the enrolled individuals will be estimated overall and by relevant factors (recruitment channel, type of advertisement) using 90% credible regions obtained by Jeffrey's prior method.
Recall of study recruitment advertisement type | 1 study session (1 hour)
  Analyses will be primarily descriptive to evaluate the reach and effectiveness of recruitment strategies. Key endpoints will be summarized overall and by relevant factors (ex., recruitment channel) using the appropriate descriptive statistics, with comparisons made using the Mann-Whitney U and Kruskal Wallis or Fisher's exact and Pearson chi-square tests, as appropriate.
Recall of recruitment channel | 1 study session (1 hour)
  Will include where study information/advertisement was viewed. Analyses will be primarily descriptive to evaluate the reach and effectiveness of recruitment strategies. Key endpoints will be summarized overall and by relevant factors ex., recruitment channel) using the appropriate descriptive statistics.
Completion method chosen by participants | 1 study session (1 hour)
  On campus versus off-campus

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Smith, PhD, Principal Investigator — Roswell Park
Locations (1):
- Roswell Park Comprehensive Cancer Center, Buffalo, New York, United States